CLINICAL TRIAL: NCT00909129
Title: Hepatitis C Virus Dynamic and Immune Activation in HIV-1 Coinfected Patients Treated With Pegylated Interferon Alfa-2a and Ribavirin
Brief Title: Interactions of Hepatitis C Viral (HCV) Dynamics and Immune Activation in HIV Coinfected Patients During HCV Treatment
Acronym: DICO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: The Swedish Research Council (Other Government); Hoffmann-La Roche (Industry)
Responsible Party: Annette Alaeus, Karolinska Institutet Sweden
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 03-541
Record Dates: First submitted 2009-05-15; First posted 2009-05-27 (Estimated); Last update posted 2009-05-27 (Estimated); Status verified 2009-05

CONDITIONS: Human Immunodeficiency Virus; Chronic Hepatitis C
Keywords: HIV-1; Chronic hepatitis C; Immune activation; HCV kinetics; IP-10
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Interferons; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HIV-1 HCV coinfected patients (Experimental): HIV-1 HCV coinfected patients undergoing HCV therapy
  Interventions: Drug: pegylated interferon-alpha (Pegasys); Drug: ribavirin (COPEGUS)

INTERVENTIONS:
Drug: pegylated interferon-alpha (Pegasys) — Pegylated interferon-alpha 2a 180 micrograms s.c. weekly
  Other Names: Pegasys (interferon)
Drug: ribavirin (COPEGUS) — ribavirin bid 800-1200 mg depending on HCV genotype and body weight
  Other Names: COPEGUS (RIBAVIRIN)

SUMMARY:
The purpose of this study is to investigate T-cell mediated immune responses to HIV-1 and HCV and determine how these responses are affected by HCV treatment and correlates to response. Furthermore, to study Interferon-inducible protein-10 (IP-10) dynamics during HCV treatment, and correlate this to treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 Hepatitis C coinfected adult patients
* Hepatitis C treatment naive
* Stable HIV-1 infection with or without cART
* > 300 CD4+ cell count

Exclusion Criteria:

* Decompensated liver disease
* Ongoing depression
* Ongoing drug abuse
* Other contraindications for interferon or ribavirin treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)

PRIMARY OUTCOMES:
Sustained virological response | 24 weeks end of treatment (EOT)

SECONDARY OUTCOMES:
T-cell mediated immune responses | baseline to 24 weeks EOT

CONTACTS AND LOCATIONS:
Overall Officials: Annette Alaeus, MD;PhD, Principal Investigator — Infectious Diseases Unit, Dept of Medicine Solna, Karolinska Institutet Stockholm
Locations (1):
- Karolinska University Hospital Solna, Stockholm, Sweden

REFERENCES:
- [Result] Gonzalez VD, Falconer K, Michaelsson J, Moll M, Reichard O, Alaeus A, Sandberg JK. Expansion of CD56- NK cells in chronic HCV/HIV-1 co-infection: reversion by antiviral treatment with pegylated IFNalpha and ribavirin. Clin Immunol. 2008 Jul;128(1):46-56. doi: 10.1016/j.clim.2008.03.521. Epub 2008 May 20. PMID 18495540
- [Derived] Falconer K, Askarieh G, Weis N, Hellstrand K, Alaeus A, Lagging M. IP-10 predicts the first phase decline of HCV RNA and overall viral response to therapy in patients co-infected with chronic hepatitis C virus infection and HIV. Scand J Infect Dis. 2010 Dec;42(11-12):896-901. doi: 10.3109/00365548.2010.498019. Epub 2010 Jul 7. PMID 20608766